CLINICAL TRIAL: NCT06878404
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of JNJ-77242113 for the Treatment of Biologic-naïve Participants With Active Psoriatic Arthritis
Brief Title: A Study to Evaluate the Efficacy and Safety of JNJ-77242113 (Icotrokinra) in Biologic-naïve Participants With Active Psoriatic Arthritis
Acronym: ICONIC-PsA 1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 77242113PSA3001; 77242113PSA3001 (Other: Janssen Research & Development, LLC); 2023-509239-19-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-03-13; First posted 2025-03-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group I: Icotrokinra Dose 1 (Experimental): Participants will receive icotrokinra dose 1. Participants who continue into a long term extension (LTE) will continue to receive icotrokinra dose 1.
  Interventions: Drug: Icotrokinra
- Group II: Icotrokinra Dose 2 (Experimental): Participants will receive icotrokinra dose 2. Participants who continue into a LTE will continue to receive icotrokinra dose 2.
  Interventions: Drug: Icotrokinra
- Group III: Placebo (Placebo Comparator): Participants will receive placebo matched to icotrokinra and will cross over to receive icotrokinra dose 1 or dose 2. Participants who continue into the LTE will continue to receive icotrokinra dose 1 or dose 2.
  Interventions: Drug: Icotrokinra; Drug: Placebo
- Group IV: Active Reference Comparator (Active Comparator): Participants will receive active reference drug. Participants who continue into a LTE will cross-over to receive icotrokinra dose 1 or dose 2.
  Interventions: Drug: Icotrokinra; Drug: Active reference comparator

INTERVENTIONS:
Drug: Icotrokinra — Icotrokinra will be administered.
  Other Names: JNJ-77242113
Drug: Placebo — Placebo will be administered.
  Arms: Group III: Placebo
Drug: Active reference comparator — Active reference drug will be administered.
  Arms: Group IV: Active Reference Comparator

SUMMARY:
The purpose of this study is to evaluate the efficacy of icotrokinra compared to placebo in participants with active psoriatic arthritis (PsA) by assessing the reduction in signs and symptoms of PsA.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of psoriatic arthritis (PsA) for at least 3 months before the first administration of study intervention and meet classification criteria for psoriatic arthritis (CASPAR) at screening
* Have active PsA as defined by: (a) At least 3 swollen joints and at least 3 tender joints at screening and at baseline (b) C-reactive protein (CRP) greater than or equal to (>=) 0.1 milligrams per deciliter (mg/dL) at screening from the central laboratory
* Have at least 1 of the PsA subsets: distal interphalangeal joint involvement, polyarticular arthritis with absence of rheumatoid nodules, arthritis mutilans, asymmetric peripheral arthritis, or spondylitis with peripheral arthritis
* Have active plaque psoriasis with at least one psoriatic plaque of >= 2 cm diameter or nail changes consistent with psoriasis
* A female participant of childbearing potential must have a negative highly sensitive serum pregnancy test (Beta-hCG) at screening and a negative urine pregnancy test at Week 0 prior to administration of study intervention

Exclusion Criteria:

* Has previously received any biologic disease-modifying antirheumatic drugs (DMARDs) for PsA or psoriasis
* Has a history or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic (with the exception of PsA), psychiatric, genitourinary, or metabolic disturbances
* Has known allergies, hypersensitivity, or intolerance to icotrokinra or its excipients
* Has other inflammatory diseases that might confound the evaluations of benefit of icotrokinra therapy, including but not limited to rheumatoid arthritis (RA), systemic lupus erythematosus, or lyme disease
* Participants with fibromyalgia or osteoarthritis symptoms that, in the investigator's opinion, would have potential to interfere with efficacy assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-05-27 (Estimated); Study Completion 2028-11-21 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants who Achieve an American College of Rheumatology (ACR) ACR 20 Response at Week 16 | Week 16
  The ACR 20 responders are participants with an improvement of greater than or equal to (>=) 20 percent (%) from baseline in both the tender and swollen joint count and in at least 3 of the 5 assessments (patient's assessment of pain visual analog scale (VAS), patient's global assessment of disease activity VAS scale, physician's global assessment of disease activity VAS scale, health assessment questionnaire and C-reactive protein).

SECONDARY OUTCOMES:
Proportion of Participants Who Achieve Psoriatic Area and Severity Index (PASI) 75 Response at Week 16 Among Participants with Baseline Body Surface Area (BSA) Greater Than Equal to (>=) 3 Percent (%) and an IGA Score of >=2 at Baseline | Week 16
  The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 75 response represents participants who achieved at least a 75 percent improvement from baseline in the PASI score.
Proportion of Participants Who Achieve PASI 90 Response at Week 16 Among Participants with Baseline BSA >=3% and an IGA Score of >=2 at Baseline | Week 16
  The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response represents participants who achieved at least a 90 percent improvement from baseline in the PASI score.
Proportion of Participants Who Achieve PASI 100 Response at Week 16 Among Participants with Baseline BSA >=3% and an IGA Score of >=2 at Baseline | Week 16
  The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 100 response represents participants who achieved at least a 100 percent improvement from baseline in the PASI score.
Proportion of Participants with an Investigator Global Assessment (IGA) Psoriasis Score of 0 or 1 And >=2 Grade Improvement From Baseline at Week 16 Among Participants with Baseline BSA >=3% and an IGA Score of >=2 at Baseline | Week 16
  Proportion of participants with an IGA psoriasis score of 0 or 1 and >=2 grade improvement from baseline at week 16 among participants with >=3% BSA and an IGA score of >=2 at baseline will be reported. The IGA documents the investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling, each using a 5-point scale: using 0 (no evidence), 1 (minimal), 2 (mild), 3 (moderate), and 4 (severe) scale. The IGA score of psoriasis is based upon the average of induration, erythema, and scaling scores. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Proportion of Participants who Achieve an ACR 50 Response at Week 16 | Week 16
  The ACR 50 responders are participants with an improvement of >= 50 % from baseline in both the tender and swollen joint count and in at least 3 of the 5 assessments (patient's assessment of pain VAS, patient's global assessment of disease activity VAS scale, physician's global assessment of disease activity VAS scale, health assessment questionnaire and C-reactive protein).
Proportion of Participants who Achieve an ACR 70 Response at Week 16 | Week 16
  The ACR 70 responders are participants with an improvement of >= 70 % from baseline in both the tender and swollen joint count and in at least 3 of the 5 assessments (patient's assessment of pain VAS, patient's global assessment of disease activity VAS scale, Physician's global assessment of disease activity VAS scale, health assessment questionnaire and C-reactive protein).
Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score At Week 16 | From Baseline to Week 16
  The HAQ-DI score consists of questions referring to 8 categories: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Responses in each functional area are scored from 0 to 3 (0=no difficulty and 3=inability to perform a task in that area). Overall score is computed as the sum of domain scores and divided by the number of domains answered. Total possible score range is 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Changes From Baseline in 36-Item Short Form Survey (SF-36) Physical Component Summary (PCS) Score at Week 16 | From Baseline to Week 16
  SF-36 is a standardized survey evaluating 8 aspects of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a domain is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Score from physical function, role physical, bodily pain, and general health domains are averaged to calculate PCS. Total score range for PCS is 0-100 (100=highest level of physical functioning).
Proportion of Participants With Resolution of Enthesitis at Week 16 Among Those With Enthesitis at Baseline | Week 16
  Enthesitis will be assessed using the Leeds Enthesitis Index (LEI). The LEI was developed to assess enthesitis in participants with PsA, and evaluates the presence (score of 1) or absence of pain (score of 0) by applying local pressure to lateral elbow epicondyle, left and right, medial femoral condyle, left and right, and achilles tendon insertion, left and right. LEI scores ranging from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness). Resolution is defined as participants have enteritis (LEI score >0) at baseline and no enthesis (LEO score =0) at the visit (week 16).
Change From Baseline in Enthesitis Score (LEI) at Week 16 in Participants With Enthesitis at Baseline | From Baseline to Week 16
  Enthesitis will be assessed using the LEI. The LEI was developed to assess enthesitis in participants with PsA, and evaluates the presence (score of 1) or absence of pain (score of 0) by applying local pressure to Lateral elbow epicondyle, left and right, Medial femoral condyle, left and right, and Achilles tendon insertion, left and right. LEI total scores ranging from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness).
Proportion of Participants With Resolution of Dactylitis at Week 16 Among Those With Dactylitis at Baseline | Week 16
  Dactylitis is characterized by swelling of the entire finger or toe. The severity of dactylitis is scored on a scale of 0-3, where 0=tenderness and 3=extreme tenderness in each digit of the hands and feet. The range of total dactylitis scores for a participant is 0-60. Higher score indicates greater degree of tenderness. Resolution is defined as participants have dactylitis (score >0) at baseline and no dactylitis (score =0) at the visit (week 16).
Change From Baseline in Dactylitis Score at Week 16 in Participants With Dactylitis at Baseline | From Baseline to Week 16
  Dactylitis is characterized by swelling of the entire finger or toe. The severity of dactylitis is scored on a scale of 0-3, where 0=tenderness and 3=extreme tenderness in each digit of the hands and feet. The range of total dactylitis scores for a participant is 0-60. Higher score indicates greater degree of tenderness.
Proportion of Participants who Achieve Minimal Disease Activity (MDA) at Week 16 | Week 16
  MDA criteria are a composite of 7 outcome measures used in PsA. Participants are classified as achieving MDA if they fulfill 5 of 7 outcome measures: tender joint count less than or equal to (<=) 1; swollen joint count <= 1; psoriasis activity and severity index <= 1 or body surface area <= 3; patient pain VAS score of <= 15; patient global disease activity VAS (arthritis and psoriasis) score of <= 20; health assessment questionnaire (HAQ) score <= 0.5; and tender entheseal points <= 1.
Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Week 16 | From Baseline to Week 16
  The FACIT-fatigue is a self-administered, 13-item questionnaire measuring items on tiredness, weakness, and difficulty conducting usual activities due to fatigue. Responses to all items are rated on a 5-point likert response scale ranging from 0 "not at all" to 4 "very much." The total score ranges from 0 to 52, with higher values indicating less fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (155):
- United States (9):
  - Arthritis and Rheumatism Associates ARA Jonesboro, Jonesboro, Arkansas
  - Omega Research Consultants, DeBary, Florida
  - Integral Rheumatology And Immunology Specialists, Plantation, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Willow Rheumatology and Wellness PLLC, Willowbrook, Illinois
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Arthritis and Rheumatology Research Institute, Allen, Texas
  - Naiara Alvarez MD Integrative Rheumatology of South TX, Harlingen, Texas
- Argentina (8):
  - Cosultorios Reumatologógicos Pampa, Buenos Aires
  - Mindout Research, Buenos Aires
  - Hospital Central Militar Cirujano Mayor Dr Cosme Argerich, Buenos Aires
  - Arsema, Ciudad de Buenos Aires
  - Centro Medico Privado de Reumatologia Tucuman, Ciudad de San Miguel de Tucuman
  - Consultora Integral de Salud SRL, Córdoba
  - MR Medicina Reumatologica, San Fernando
  - Instituto Medico De Alta Complejidad (IMAC), San Isidro
- Australia (5):
  - Ipswich Hospital, Ipswich
  - Rheumatology Research Unit, Maroochydore
  - BJC Health, Parramatta
  - Queen Elizabeth Hospital, South Woodville
  - Royal Darwin Hospital, Tiwi
- Bulgaria (4):
  - MC Medtech Services Ltd, Haskovo
  - Exacta Medica, Pleven
  - Medical Center Artmed, Plovdiv
  - Medical Center Teodora, Rousse
- China (23):
  - Peking University Third Hospital, Beijing
  - Beijing Tong Ren Hospital Capital Medical University, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - West China Hospital Sichuan University, Chengdu
  - Sichuan Provincial Peoples Hospital, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Nanfang Hospital of Southern Medical Hospital, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Linyi City People Hospital, Linyi
  - Jiangxi Provincial Peoples Hospital, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Affiliated Hospital of Nantong University, Nantong
  - Pingxiang People's Hospital, Pingxiang
  - Huashan Hospital Fudan University, Shanghai
  - Shanghai skin disease hospital, Shanghai
  - Shenzhen People s Hospital, Shenzhen
  - The Third Hospital of Hebei Medical University, Shijiazhuang
  - Second Affiliated Hospital of Soochow University, Suzhou
  - Shanxi Bethune Hospital, Taiyuan
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Affiliated Hospital of Jiangsu University, Zhenjiang
- Czechia (13):
  - Revmatologie s r o, Brno
  - Revmacentrum MUDr Mostera s r o, Brno-Židenice
  - RHEUMA s r o, Břeclav
  - Revmatologicka ambulance, Fryštát
  - L K N Arthrocentrum, Hlučín
  - CCR Ostrava S R O, Ostrava
  - MUDr Rosypalova s r o, Ostrava
  - Revmatologicky ustav, Prague
  - Revmatologicka ambulance, Prague
  - Thomayerova nemocnice, Prague
  - FN Motol, Prague
  - Medical Plus S R O, Uherské Hradiště
  - PV Medical S R O, Zlín
- Denmark (6):
  - Aarhus University Hospital, Aarhus N
  - Sydvestjysk Sygehus, Esbjerg
  - Frederiksberg Hospital, Frederiksberg
  - Regionshospitalet Godstrup, Herning
  - Svendborg Hospital Odense University Hospital, Svendborg
  - Vejle Sygehus, Vejle
- Germany (10):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Charite Universitaetsmedizin Berlin, Berlin
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - Medizinische Fakultat der Albert Ludwigs Universitat Freiburg, Freiburg im Breisgau
  - Hamburger Rheuma Forschungszentrum II, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
  - Studienzentrum Dr Schwarz Germany, Langenau
  - Johannes Wesling Klinikum Minden, Minden
  - Universitatsklinikum Tubingen, Tübingen
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Hungary (12):
  - Betegapolo Irgalmas Rend Budai Irgalmasrendi Korhaz, Budapest
  - Revita Kft, Budapest
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Qualiclinic Kft, Budapest
  - Synexus Magyarorszag Kft, Budapest
  - Uno Medical Trials Ltd., Budapest
  - University of Debrecen, Debrecen
  - Bekes Varmegyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - Obudai Egeszsegugyi Centrum Kft, Kaposvár
  - University of Szeged, Szeged
  - MAV Korhaz es Rendelointezet, Szolnok
  - Vital Medical Center Orvosi es Fogaszati Kozpont, Veszprém
- India (10):
  - Marengo Cims Hospital, Ahmedabad
  - Apollo Hospitals, Bhubaneswar
  - Nizams Institute of Medical Sciences, Hyderabad
  - Apollo Multispeciality Hospital Ltd, Kolkata
  - Kokilaben Dhirubhai Ambani Hsp And Med Research Inst, Mumbai
  - JSS Hospital, Mysuru
  - All India Institute of Medical Sciences, New Delhi
  - Indraprastha Apollo Hospital, New Delhi
  - Fortis Hospital, Noida
  - SIDS Hospital & Research Centre, Surat
- Japan (10):
  - Fukuoka University Hospital, Fukuoka
  - Teikyo University Hospital, Itabashi Ku
  - Kagawa University Hospital, Kita Gun
  - Nagoya City University Hospital, Nagoya
  - Public Interest Incorporated Foundation Nipoon Life Saiseikai Nippon Life Hospital, Osaka
  - Maeshima Rheumatology Clinic, Ōita
  - Sasebo Chuo Hospital, Sasebo
  - Tohoku University Hospital, Sendai
  - Kyorin University Hospital, Tokyo
  - Mie University Hospital, Tsu
- Poland (20):
  - Osteo Medic S C Artur Racewicz Jerzy Supronik, Bialystok
  - Specderm Poznanska sp j, Bialystok
  - ClinicMed Daniluk Nowak Spolka Komandytowa, Bialystok
  - Szpital Uniwersytecki Nr 2 w Bydgoszczy, Bydgoszcz
  - Ambulatorium sp. z o.o., Elblag
  - Centrum Kliniczno Badawcze, Elblag
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Malopolskie Badania Kliniczne Sp z o o, Krakow
  - Specjalistyczny gabinet dermatologiczny Aplikacyjno Badawczy Marek Brzewski Pawel Brzewski Spolka Cywilna, Krakow
  - Centrum Medyczne All Med, Krakow
  - Pratia MCM Krakow, Krakow
  - Dermed Centrum Medyczne Sp z o o, Lodz
  - Zespol Poradni Specjalistycznych Reumed Filia nr 1, Lublin
  - NZOZ Lecznica MAK MED S C, Nadarzyn
  - Etyka Osrodek Badan Klinicznych, Olsztyn
  - MICS Centrum Medyczne Torun, Torun
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Centrum Medyczne Reuma Park, Warsaw
  - DermMedica Sp z o o, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
- Spain (12):
  - Hosp Univ A Coruna, A Coruña
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Clinic de Barcelona, Barcelona
  - Hosp Reina Sofia, Córdoba
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Macarena, Seville
  - Hosp. Infanta Luisa, Seville
  - Hosp. Quiron Sagrado Corazon, Seville
  - Hosp. Virgen Del Rocio, Seville
- Taiwan (6):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center Yong Kang, Tainan
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital Hsin Chu Branch, Taoyuan District
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Thailand (6):
  - Phramongkutklao Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Saraburi Hospital, Changwat Sara Buri
  - Phra Nakhon Si Ayutthaya Hospital, Phra Nakhon Si Ayutthaya
  - Songklanagarind hospital, Songkhla

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency